CLINICAL TRIAL: NCT01307215
Title: Lumbar Transversus Abdominal Plane (TAP) Block: Does Volume Make a Difference?
Brief Title: TAP Block: Does Volume Make a Difference?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 10-3436
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2011-05

CONDITIONS: Post-operative Pain
Keywords: TAP block; incision pain; total hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 20mLs of 0.5% ropivacaine per side (Experimental)
  Interventions: Drug: Ropivacaine
- 30mLs of 0.33% ropivacaine per side (Experimental)
  Interventions: Drug: Ropivacaine
- 40mLs of 0.25% ropivacaine per side (Experimental)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — 20mLs of 0.5%
  Other Names: naropeine; naropin
  Arms: 20mLs of 0.5% ropivacaine per side
Drug: Ropivacaine — 30mLs of 0.33%
  Other Names: naropeine; naropin
  Arms: 30mLs of 0.33% ropivacaine per side
Drug: Ropivacaine — 40mLs of 0.25%
  Other Names: naropeine; naropin
  Arms: 40mLs of 0.25% ropivacaine per side

SUMMARY:
Patients who have abdominal surgery will experience pain from the incision. The lumbar TAP block is a procedure used to reach the nerve endings in the abdominal wall so that there is a reduction in pain after surgery. Using ultrasound guidance, a solution of ropivacaine will be injected after surgery. The aim of this study is to determine the effect of changes in the volume of the injection.

DETAILED DESCRIPTION:
Pain from a surgical incision happens in most patients. During the perioperative period, the use of the TAP block has been shown to reduce pain scores, opioid consumption and sedation scores. Also, there is a trend towards a reduction of post-operative nausea and vomiting. The aim of the block is to reach the distal nerve endings of the abdominal wall from T6 to L1 dermatomes using ultrasound guidance with a single shot of ropivacaine at different volumes. Currently, there is consensus about optimal procedure-specific volumes and local anesthetic concentrations for lumbar TAP blocks. This is a pilot study and the purpose being is it feasible to do a large scale clinical study to determine the influence of increasing the local anesthetic volume.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* total abdominal hysterectomy
* capable of completing informed consent
* no previous chronic opioid use
* no previous abdominal wall surgeries

Exclusion Criteria:

* patient refusal
* contraindication to regional anesthesia: coagulopathy, anticoagulant use, bleeding disorders,
* local or systemic infection
* local anesthetic allergy
* BMI>35

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of a large scale clinical study to determine the influence on increasing the local anesthetic volume. | 6 month
  This will be shown as a number and a percenttage of patients recruited and randomized.

SECONDARY OUTCOMES:
Using ice and pinprick, determine the dermatomal block distribution at 2,6,12,24 and 48 hours post block. | 48 hours
  The assessor will measure the extend of the block distribution at the various time intervals.
Pain scores at 2,6,12,24, and 48 hours post-block. | 48 hours
  Using a visual analog scale, patient pain scores will be assessed.
Patient-controlled analgesia opioid requirements at 2,6,12,24 and 48 post-block. | 48 hours
  Record drug consumption at the time intervals
Incidence of post-operative nausea and vomiting at 2,6,12,24, and 48 hours. | 48 hours
Block failure rate. | 48 hours
  Block failure rate is defined as the lack of any sensory block following the TAP block.
Patient's overall satisfaction. | 48 hours
  Using a LIKERT score, patient satisfaction will be measured.
Discharge time from PACU. | 24 hours
  The time in which the patient is discharged from the recovery room.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Forero, MD, Principal Investigator — McMaster University/St. Joseph's Healthcare
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Petersen PL, Mathiesen O, Torup H, Dahl JB. The transversus abdominis plane block: a valuable option for postoperative analgesia? A topical review. Acta Anaesthesiol Scand. 2010 May;54(5):529-35. doi: 10.1111/j.1399-6576.2010.02215.x. Epub 2010 Feb 17. PMID 20175754
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Derived] Forero M, Heikkila A, Paul JE, Cheng J, Thabane L. Lumbar transversus abdominis plane block: the role of local anesthetic volume and concentration-a pilot, prospective, randomized, controlled trial. Pilot Feasibility Stud. 2015 Mar 25;1:10. doi: 10.1186/s40814-015-0002-6. eCollection 2015. PMID 27965789